CLINICAL TRIAL: NCT01430923
Title: Randomized,Active Comparator-Controlled,Three Months,Open Label Clinical Trial to Compare Efficacy and Safety of Refrigeration-Free Latanoprost (0.005%) and Latanoprost (0.005%) Stored at Refrigeration Temperature in Patients With OAG or OHT
Brief Title: Clinical Evaluation of Safety and Efficacy of Refrigeration Free Latanoprost
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aurolab (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LATANOPROST/CIP/002/2011
Record Dates: First submitted 2011-09-07; First posted 2011-09-09 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
Keywords: Refrigeration free latanoprost
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Refrigeration free Latanoprost (Experimental): Latanoprost refrigeration free formulation as per randomization schedule.
  Interventions: Drug: refrigeration free latanoprost
- latanoprost 2-8˚ C (Active Comparator): latanoprost stored at 2-8˚ C
  Interventions: Drug: latanoprost eye drops

INTERVENTIONS:
Drug: refrigeration free latanoprost — latanoprost Eye drops 0.005% once daily, 3 months
  Other Names: Auroprost RT
  Arms: Refrigeration free Latanoprost
Drug: latanoprost eye drops — latanoprost eye drops 0.005% w/v, once daily, 3 months
  Other Names: Auroprost
  Arms: latanoprost 2-8˚ C

SUMMARY:
The purpose of this study is to:

* To evaluate the efficacy of Refrigeration-Free Latanoprost compared to Latanoprost stored at refrigeration temperature with respect to the diurnal intraocular pressure (IOP) change from baseline after 3 months of therapy in patients with open-angle glaucoma (OAG) or ocular hypertension.
* To evaluate the safety and tolerability of Refrigeration-Free Latanoprost in patients with open-angle glaucoma (OAG) or ocular hypertension.

DETAILED DESCRIPTION:
Latanoprost refrigeration free formulation is developed to overcome difficulties on storing drugs at 2-8˚ C in consumer end and also to avoid risk during transition. This formulation has the best solubilizing agent cyclodextrin to increase the solubility and stability of latanoprost API. To find out the efficacy and safety due to this additional excipient in this formulation rather than the cold storage product the investigators have to perform clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patient between 18 and 80 years of age
* Newly diagnosed Primary Open-Angle Glaucoma, Pigmentary Glaucoma, Pseudoexfoliation, or Ocular hypertension.
* Patient has a mean (or median) IOP of 24 and 36 mmHg in at least one eye
* Patient has a best corrected ETDRS visual acuity score of +0.6 logMAR (Snellen equivalent of 20/80) or better in each eye.
* Patient should have the access / ability to refrigerate study drug.
* Residence with 60 kms of Madurai

Exclusion Criteria:

* Patient has a mean (or median) IOP >36 mmHg in either eye at the Screening Visit.
* Patient has a history of or current abnormal corneal sensation or any abnormality in either eye preventing reliable Goldmann applanation tonometry
* Pupil in either eye that will not dilate sufficiently for adequate evaluation of the retina
* Patient has a history of retinal detachment, proliferative diabetic retinopathy, or any retinal disease in either eye that may be progressive during the study
* Patient who has significant ocular symptoms or signs such as photophobia, flashes or streaks of light, metamorphopsia, diplopia, or transient loss of vision in either eye.
* Patient has had intraocular surgery (e.g., cataract extraction) in either eye within 4months prior to Screening visit.
* Patient is aphakic or has, in the judgement of the investigator, risk for ocular inflammation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-05 (Actual); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure | 3 months
  to evalate the change in intraocular pressure from baseline to end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Manju R Pillai, MBBS.,, Principal Investigator — Araving Eye Hospital
Locations (1):
- Aravind Eye hospital, Madurai, Tamil Nadu, India